CLINICAL TRIAL: NCT04229888
Title: Meibomian Gland Dysfunction Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Anna Tichenor, Assistant Scientist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1908329543
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
Keywords: dry eye; meibomian gland dysfunction; lipiflow
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: All subjects will receive first treatment and then second treatment. The eye receiving treatment will be randomly selected. The same eye will receive both treatments.
Masking Description: Outcomes assessor blinded to visit schedule. Participants masked to invalidity of sham treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subject Treatment (Experimental): All subjects will receive light based (sham) treatment, then all subjects will receive LipiFlow treatment.
  Interventions: Device: LipiFlow; Device: Light Based (Sham) Treatment

INTERVENTIONS:
Device: LipiFlow — Medical device that applies a combination of heat and pressure to the inner eyelid to remove gland obstructions and stagnant gland content
  Other Names: Johnson & Johnson
Device: Light Based (Sham) Treatment — A light based (sham) treatment will be used to compare effectiveness to the LipiFlow treatment.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of treatments for Meibomian Gland Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* evidence of meibomian gland obstruction in both eyes
* dry eye symptoms per DEQ-5

Exclusion Criteria:

* active ocular infection
* previous LipiFlow treatment
* beginning new oral or other systemic medications within prior 3 months
* beginning new or changing dosages of ocular medications within prior 3 months
* previous ocular surgery, trauma, herpes, recurrent inflammation, punctal plugs in prior 3 months
* habitual contact lens wear in prior 3 months
* women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Optometry, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 subjects total were enrolled which is less than what was expected (15) due to time constraints
Period: Overall Study
Arm/Group | Subject Treatment
Started (All 14 subjects total received both treatments) | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subject Treatment: All subjects will receive light based treatment, then all subjects will receive LipiFlow treatment.
Arm/Group | Subject Treatment
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.57 (16.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Dry Eye Questionnaire 5 (DEQ-5) Score
Description: DEQ5 total score ranges from 0-22 with the higher scores indicating increased dry eye.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Subjects Treatment Light Based (Sham): All subjects will receive light based (sham) treatment.
  Light Based Treatment: A light based (sham) treatment will be used to compare effectiveness to the LipiFlow treatment.
- Subjects Treatment LipiFlow: All subjects will receive LipiFlow treatment.
  LipiFlow: Medical device that applies a combination of heat and pressure to the inner eyelid to remove gland obstructions and stagnant gland content
Arm/Group | Subjects Treatment Light Based (Sham) | Subjects Treatment LipiFlow
Number analyzed (Participants) | 14 | 14
score on a scale | 11.8 (3.9) | 11.8 (4.4)
Statistical Analysis 1: Comparison: Subjects Treatment Light Based (Sham) vs Subjects Treatment LipiFlow; Test type: Non-Inferiority — To establish non-inferiority of the treatment effect on the primary outcome change in DEQ-5 score, the upper bound of the two-sided 95% confidence interval on mean difference between the light based (sham) treatment and Lipiflow treatment were compared against a non-inferiority margin M=6 representing the largest clinically acceptable difference based on historical data; p = 0.02, ANOVA

2. Secondary Outcome: Meibomian Gland Score
Description: Meibomian glands evaluated on the lower eyelid using meibomian gland evaluator. 5 glands in 3 regions (nasal, central, temporal) evaluated and scored from 0 to 4 for a max score of 60 in each eye. (MGS scale 0 = clear, 1 = cloudy, 2 = granular, 3 = pastelike, 4 = obstruction)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Subjects Treatment Light Based (Sham): All subjects will receive light based (sham) treatment.
  Light Based Treatment: A light based treatment will be used to compare effectiveness to the LipiFlow treatment.
Arm/Group | Subjects Treatment Light Based (Sham) | Subjects Treatment LipiFlow
Number analyzed (Participants) | 14 | 14
score on a scale | 53.2 (7.9) | 52.6 (7.9)
Statistical Analysis 1: Comparison: Subjects Treatment Light Based (Sham) vs Subjects Treatment LipiFlow; Test type: Non-Inferiority — To establish non-inferiority of the treatment effect on the primary outcome change in MG score, the upper bound of the two-sided 95% confidence interval on mean difference between the light based (sham) treatment and Lipiflow treatment were compared against a non-inferiority margin M= 1 representing the largest clinically acceptable difference based on historical data; p = 0.07, ANOVA

3. Secondary Outcome: Tear Break-Up Time (TBUT)
Description: Tear break-up time (defined as the time required for dry spots to appear on the surface of the eye after blinking) was assessed by the examiner using a slit lamp and fluorescein strips. Fluorescein was instilled onto the patient's eye, after which the patient blinked three times, then kept the eye open. Immediately thereafter, the examiner used a stopwatch to record the time between the last blink and the first appearance of a dark spot on the cornea (formation of dry area). Three consecutive measurements were taken and averaged for actual TBUT. A positive change value represents a lengthening in the tear break-up time and greater comfort.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Subjects Treatment Light Based (Sham) | Subjects Treatment LipiFlow
Number analyzed (Participants) | 14 | 14
seconds | 7.11 (9.09) | 5.62 (6.77)
Statistical Analysis 1: Comparison: Subjects Treatment Light Based (Sham) vs Subjects Treatment LipiFlow; Test type: Non-Inferiority — To establish non-inferiority of the treatment effect on the primary outcome change in TBUT, the upper bound of the two-sided 95% confidence interval on mean difference between the light based (sham) treatment and Lipiflow treatment were compared against a non-inferiority margin M=6 representing the largest clinically acceptable difference based on historical data; p = 0.66, ANOVA

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Light Based (Sham) Treatment; LipiFlow Treatment: All subjects will receive light based (sham) treatment, then all subjects will receive LipiFlow treatment.
Arm/Group | Light Based (Sham) Treatment | LipiFlow Treatment
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT04229888/Prot_SAP_000.pdf